CLINICAL TRIAL: NCT03165331
Title: Online Psychosocial Support for Young People Distressed by Appearance-altering Conditions: A Randomised Control Trial (RCT)
Brief Title: Online Psychosocial Support for Young People With a Visible Difference: A Randomised Control Study
Acronym: UNGFaceIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Oslo University Hospital (Other)
Collaborators: Centre for Appearance Research, University of the West of England, UK (Unknown)
Responsible Party: Principal Investigator, Kristin Billaud Feragen, Research Coordinator at the Centre for Rare Disorders, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015/2440-4
Record Dates: First submitted 2017-05-23; First posted 2017-05-24 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Skin Condition; Cleft Lip and Palate; Burns; Other Conditions Leading to a Visible Difference; Craniofacial Abnormalities
MeSH Terms: conditions — Skin Diseases; Cleft Lip; Burns; Craniofacial Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Other): The intervention group will go through the intervention programme (Ung Face IT) after T1 and randomisation. Programme takes 7 weeks to complete + Treatment as usual (local health care services). Questionnaires after the 7 weeks (T2) and after three months (T3) and 6 months (T4).
  Interventions: Other: Ung Face IT
- Control group (Other): Treatment as usual for three months after T1 and randomisation, with local health care support if needed. Questionnaires at T2 and T3 before participants are given access to the intervention (Ung Face IT) after three months. Questionnaire at T4 (post-intervention).
  Interventions: Other: Ung Face IT

INTERVENTIONS:
Other: Ung Face IT — Ung Face IT is an online intervention tool (programme) that provides easy access to specialist advice and support via a home computer/tablet, using illustrations, information, videos, and interactive activities, and a discussion forum for participants only (supervised by the research team). Through these tools, it provides advice and teaches coping skills based on cognitive behavioural therapy and social interaction skills training.
  Other Names: English name: Young People Face IT (YP Face IT)

SUMMARY:
A visible difference can have a profound impact in a society with a massive emphasis on appearance and "looks". A vulnerable group is adolescents with a condition affecting their appearance as a result of injuries (burns, accidents), treatment (cancer), skin conditions or congenital anomalies (birthmarks, craniofacial conditions). Research has identified potential psychological difficulties, which, if not addressed, can lead to anxiety, depression, and eating disorders.

In addition to medical treatment options, aiming at diminishing a difference that may be visible to others, young people with appearance concerns also need self-management skills. However, evidence-based interventions are scarce and specialised psychological treatment is difficult to reach.

The Centre for Appearance Research (Bristol, UK) has developed an online intervention for adolescents, now translated into Norwegian (www.ungfaceit.no). UNG Face IT provides easy access to specialist advice and support via a home computer, using information, videos, and interactive activities. It provides advice, teaches coping and social skills, strengthening psychological adjustment to a visible difference.

A systematic evaluation of the Norwegian version is needed. UNG Face IT could potentially address unmet needs, provide a cost-effective tool to reduce the need for "face-to-face" psychological and surgical/medical services, and contribute to make online health care available for young people with a visible difference.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-17 with an appearance-altering condition, and experiencing appearance-related distress, teasing, or bullying
* Access to a home computer/tablet and internet
* Reading level > 12 years of age. Audio recordings for all written text available on the website for those who may struggle with reading
* Normal/corrected-to-normal vision

Exclusion Criteria:

* Clinical depression, psychosis, eating disorder (alternative support necessary)
* Post-traumatic stress disorder (PTSD) or within 12 months of traumatic injury (alternative support necessary)
* Learning disability that would impede understanding of the programme's content
* Currently receiving psychological intervention

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 130 (Estimated)
Dates: Start 2016-04-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Body Esteem Scale (BES) | 6 months
  Includes three subscales, only the subscale BE_Appearance used in this study. Measures general feelings about appearance.

SECONDARY OUTCOMES:
Life Engagement Scale (LES) | 6 months
  Social experiences and social engagement (10 items)
Perceived Stigmatisation Questionnaire | 6 months
  Three subscales: Absence of friendly behaviour, confused and staring behaviour, and hostile behaviour by others. These communicate social acceptance, social discomfort, and social rejection respectively.
Harter's Self-Perception Profile for Adolescents | 6 months
  Two subscales are used: Romantic concerns and general self-esteem
EQ-5D-5L | 6 months
  Indicator of the impact of UNG Face IT on Health related quality of life and to provide Health economic data
Resource Use Questionnaire (Parents) | 6 months
  Assessing time out of School, use of Health care Resources and expenses in relation to the child's condition.

CONTACTS AND LOCATIONS:
Overall Officials: Olve Moldestad, PhD, Study Director — Centre Director
Locations (1):
- Centre for Rare Disorders, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Data from the UK and Nethelands will be shared anonymously with the Norwegian Research team. No Norwegian data will be shared with international collaborators.

REFERENCES:
- [Derived] Zelihic D, Feragen KJB, Pripp AH, Nordgreen T, Williamson H, Kling J. Predictors of Adolescents' Response to a Web-Based Intervention to Improve Psychosocial Adjustment to Having an Appearance-Affecting Condition (Young Person's Face IT): Prospective Study. JMIR Form Res. 2023 Jan 18;7:e35669. doi: 10.2196/35669. PMID 36652281
- [Derived] Millgard M, Feragen KB, Ullmann Miller J, Arfa S, Williamson H, Kling J. Adolescents and parents' perception of Young Person's Face IT: An online intervention for adolescents struggling with conditions affecting their appearance. Digit Health. 2022 Dec 25;8:20552076221147110. doi: 10.1177/20552076221147110. eCollection 2022 Jan-Dec. PMID 36601286